CLINICAL TRIAL: NCT00013299
Title: Clinical Trials of Footwear in Patients With Diabetes-Study Arm 2,3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A2443R
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2001-01

CONDITIONS: Diabetic Foot Ulcers
Keywords: Foot ulcers, amputation prevention, diabetes, footwear, insoles
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Diabetes Mellitus

INTERVENTIONS:
Device: Prevention of Diabetic Ulcers

SUMMARY:
This is a randomized clinical trial to: (1) Determine the extent to which custom made study shoes will reduce the incidence of reulceration in diabetic individuals with prior history of foot ulcers, and (2) Estimate costs of ulcer prevention using these strategies.

DETAILED DESCRIPTION:
This is a randomized clinical trial to: (1) Determine the extent to which custom made study shoes will reduce the incidence of reulceration in diabetic individuals with prior history of footulcers, and (2) Estimate costs of ulcer prevention using these strategies. Patients from the Seattle VA (n=214) and Group Health Cooperative (n=213) will be randomly assigned to one of two study arms. They are: (1) patients wearing study shoes and premolded polyurethane insoles and (2) the control group of patients wearing their own footwear.

ELIGIBILITY:
Diabetics with foot ulcerations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427
Dates: Start 2000-10; Study Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Fryer, Ph.D. Asst. Director — Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service; Wijegupta Ellepola, Program Analyst — Program Analysis and Review Section (PARS), Rehabilitation Research & Development Service
Locations (1):
- VAMC, Seattle, WA, Seattle, Washington, United States